CLINICAL TRIAL: NCT03504631
Title: Genotyping and Phenotyping of CYP2D6 as Predictor of Z-endoxifen Plasma Levels in Breast Cancer Patients on Tamoxifen Treatment
Brief Title: Genotyping and Phenotyping of CYP2D6 Breast Cancer Patients on Tamoxifen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trisakti University (Other)
Collaborators: Dharmais National Cancer Center Hospital (Other Government)
Responsible Party: Principal Investigator, Yenny Farmako, Head of Pharmacology, Trisakti University
Other Study IDs: 1001
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer Female
Keywords: tamoxifen; breast cancer; Z-endoxifen
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples from breast cancer patients treated with Z-endoxifen were drawn for analysis of genotype and phenotype of CYP2D6, as well as the plasma concentration of Z-endoxifen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients on tamoxifen: Patients currently on treatment with tamoxifen for at least 4 months.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
This study is an observational study to determine phenotype and genotype of CYP2D6 as predictors of z-endoxifen concentrations in plasma of outgoing patients treated with tamoxifen for at least 4 months

DETAILED DESCRIPTION:
Tamoxifen is an antiestrogen drug with concentration dependent properties, with z-endoxifen known as active metabolite. Until know therapeutic range for z-endoxifen to improve treatment response was not known. Variation response on tamoxifen can be cause of genetic polymorphism CYP2D6 that can be different between interindividul and ethnic.

The aim of this study is to determine phenotype and genotype of CYP2D6 as predictors of z-endoxifen concentrations in plasma of outgoing patients treated with tamoxifen for at least 4 months

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients on tamoxifen treatment for at least 4 months

Exclusion Criteria:

* Abnormalities in liver markers (AST >2.5 x ULN)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female only
Study Population: Outpatient breast cancer patients on tamoxifen treatment for at least 4 months
Sampling Method: Non-Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Genotype and phenotype of CYP2D6 | 4 months
  Number of subjects with CYP2D6 genotype and phenotype who had steady state level

SECONDARY OUTCOMES:
Z-endoxifen | 4 months
  Number of subjects with plasma levels of Z-endoxifen more than 5.9 ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Rianto Setiabudy, MD, PhD, Study Director — Indonesia University
Locations (1):
- Dharmais hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madlensky L, Natarajan L, Tchu S, Pu M, Mortimer J, Flatt SW, Nikoloff DM, Hillman G, Fontecha MR, Lawrence HJ, Parker BA, Wu AH, Pierce JP. Tamoxifen metabolite concentrations, CYP2D6 genotype, and breast cancer outcomes. Clin Pharmacol Ther. 2011 May;89(5):718-25. doi: 10.1038/clpt.2011.32. Epub 2011 Mar 23. PMID 21430657
- [Background] Jager NG, Rosing H, Schellens JH, Linn SC, Beijnen JH. Tamoxifen dose and serum concentrations of tamoxifen and six of its metabolites in routine clinical outpatient care. Breast Cancer Res Treat. 2014 Feb;143(3):477-83. doi: 10.1007/s10549-013-2826-1. Epub 2014 Jan 5. PMID 24390246
- [Background] Tamminga WJ, Wemer J, Oosterhuis B, Brakenhoff JP, Gerrits MG, de Zeeuw RA, de Leij LF, Jonkman JH. An optimized methodology for combined phenotyping and genotyping on CYP2D6 and CYP2C19. Eur J Clin Pharmacol. 2001 May;57(2):143-6. doi: 10.1007/s002280100273. PMID 11417446
- [Background] Desta Z, Ward BA, Soukhova NV, Flockhart DA. Comprehensive evaluation of tamoxifen sequential biotransformation by the human cytochrome P450 system in vitro: prominent roles for CYP3A and CYP2D6. J Pharmacol Exp Ther. 2004 Sep;310(3):1062-75. doi: 10.1124/jpet.104.065607. Epub 2004 May 24. PMID 15159443
- [Background] Fotoohi AK, Karim H, Lafolie P, Pohanka A, Ostervall J, Hatschek T, Vitols S. Pronounced Interindividual But Not Intraindividual Variation in Tamoxifen and Metabolite Levels in Plasma During Adjuvant Treatment of Women With Early Breast Cancer. Ther Drug Monit. 2016 Apr;38(2):239-45. doi: 10.1097/FTD.0000000000000257. PMID 26485084
- [Background] Hennig EE, Piatkowska M, Karczmarski J, Goryca K, Brewczynska E, Jazwiec R, Kluska A, Omiotek R, Paziewska A, Dadlez M, Ostrowski J. Limited predictive value of achieving beneficial plasma (Z)-endoxifen threshold level by CYP2D6 genotyping in tamoxifen-treated Polish women with breast cancer. BMC Cancer. 2015 Aug 1;15:570. doi: 10.1186/s12885-015-1575-4. PMID 26232141
- [Background] Antunes MV, Linden R, Santos TV, Wallemacq P, Haufroid V, Classen JF, Andreolla H, Costa N, Fontanive TO, Rosa DD. Endoxifen levels and its association with CYP2D6 genotype and phenotype: evaluation of a southern Brazilian population under tamoxifen pharmacotherapy. Ther Drug Monit. 2012 Aug;34(4):422-31. doi: 10.1097/FTD.0b013e318260b46e. PMID 22777153
- [Background] Lei L, Wang X, Wu XD, Wang Z, Chen ZH, Zheng YB, Wang XJ. Association of CYP2D6*10 (c.100C>T) polymorphisms with clinical outcome of breast cancer after tamoxifen adjuvant endocrine therapy in Chinese population. Am J Transl Res. 2016 Aug 15;8(8):3585-92. eCollection 2016. PMID 27648149
- [Background] Hawse JR, Subramaniam M, Cicek M, Wu X, Gingery A, Grygo SB, Sun Z, Pitel KS, Lingle WL, Goetz MP, Ingle JN, Spelsberg TC. Endoxifen's molecular mechanisms of action are concentration dependent and different than that of other anti-estrogens. PLoS One. 2013;8(1):e54613. doi: 10.1371/journal.pone.0054613. Epub 2013 Jan 28. PMID 23382923
- [Background] Bagheri A, Kamalidehghan B, Haghshenas M, Azadfar P, Akbari L, Sangtarash MH, Vejdandoust F, Ahmadipour F, Meng GY, Houshmand M. Prevalence of the CYP2D6*10 (C100T), *4 (G1846A), and *14 (G1758A) alleles among Iranians of different ethnicities. Drug Des Devel Ther. 2015 May 13;9:2627-34. doi: 10.2147/DDDT.S79709. eCollection 2015. PMID 25999696
- [Background] Zhou SF. Polymorphism of human cytochrome P450 2D6 and its clinical significance: Part I. Clin Pharmacokinet. 2009;48(11):689-723. doi: 10.2165/11318030-000000000-00000. PMID 19817501